CLINICAL TRIAL: NCT01211730
Title: Prospective, Randomized, Open-Label, Controlled Study to Evaluate the Safety and Efficacy of Intensive Glycemic Control on Outcomes Following Liver Transplantation
Brief Title: Study of Glycemic Control on Liver Transplantation Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Mark Molitch, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00005806
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Evidence of Liver Transplantation; Hyperglycemia; Rejection
Keywords: Liver; transplantation; Glucose; Hyperglycemia; Insulin; Rejection; Hypoglycemia
MeSH Terms: conditions — Hyperglycemia; Rejection, Psychology; Insulin Resistance; Hypoglycemia | interventions — Insulin; Insulin Glargine; Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 140 Group (Active Comparator): Insulin treatment to target blood glucose at 140 mg/dl
  Interventions: Drug: Insulin
- 180 Group (Active Comparator): Insulin treatment to target blood glucose at 180 mg/dl
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin initially as continuous infusion for first 24-48 hours followed by subcutaneous administration once subjects eating and out of intensive care unit.
  Other Names: glargine insulin; aspart insulin; Lantus insulin; Novolog insulin; Detemir insulin; Levemir insulin

SUMMARY:
Many but not all studies have shown improvement in morbidity and mortality with intensive glycemic management postoperatively. In this study, the investigators propose to determine whether improved glycemic control using intensive insulin treatment immediately postoperatively will improve outcomes in patients undergoing liver transplant using a prospective, controlled, randomized, parallel-group study design targeting two different glucose levels, 140 and 180 mg/dL.

DETAILED DESCRIPTION:
Many studies have shown improvement in morbidity and mortality with intensive glycemic management postoperatively. However, some recent studies have not been able to reproduce these benefits and have raised the issue of adverse consequences of hypoglycemia associated with intensive therapy. Our own data show an association of increased graft rejection proportional to postoperative glucose levels in patients who have undergone a liver transplant. Preliminary data suggest that this may improved by better glycemic control using the Glucose Management Service here at Northwestern.

In this study, we propose to determine whether improved glycemic control using intensive insulin treatment immediately postoperatively will improve outcomes in patients undergoing liver transplant using a prospective, controlled, randomized, parallel-group study design targeting two different glucose levels, 140 and 180 mg/dL. Postoperative glucose management with insulin will be supervised by the Glucose Management Service as is routine, with the only research aspect being the two different glucose targets and the outcome analysis with liver transplant rejection as the primary outcome and infections and hypoglycemia being the principle secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Require Liver Transplantation
2. Age 18 - 80
3. Able to give informed consent personally or via a family member who has appropriate authorization to do so if patient unconscious.
4. Expected survival following transplantation for > 1 year.
5. Glucose level over 180 mg/dL postoperatively

Exclusion Criteria:

1. Inability of patient or family member to give informed consent
2. Not expected to survive for > 1 year following liver transplantation.
3. Previous liver transplantation
4. Acute liver failure
5. Living related donor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2009-04; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Molitch, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were primarily recruited from Liver Transplant Clinic and the inpatient Liver Transplant service
Pre-assignment Details: Of 278 patients Consented, 46 died before transplant, 38 did not undergo transplant, 14 were delisted for transplant, and 16 did not enter the study for miscellaneous reasons.
Period: Overall Study
Arm/Group | 140 Group | 180 Group
Started | 82 | 82
Completed | 82 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing liver transplantation
Groups:
- Total: Total of all reporting groups
Arm/Group | 140 Group | 180 Group | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (8.0) | 56.9 (7.6) | 57.5 (7.8)
Gender [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 53 | 53 | 106
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 57 | 63 | 120
  Black | 6 | 9 | 15
  Hispanic | 15 | 7 | 22
  Asian | 1 | 1 | 2
  Unknown | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 82 | 82 | 164
body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (6.0) | 30.0 (6.6) | 30.1 (6.3)
Model for End-stage Liver DIsease (MELD) Score [Mean (Standard Deviation); unit: units on a scale] — The MELD Score uses the patient's values for serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time (INR) to predict survival. It is calculated according to the following formula: MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43.
  In interpreting the MELD Score in hospitalized patients, the 3 month mortality is:
  40 or more - 71.3% mortality 30-39 - 52.6% mortality 20-29 - 19.6% mortality 10-19 - 6.0% mortality <9 - 1.9% mortality
  units on a scale | 27.3 (9.4) | 28.2 (7.6) | 27.8 (8.6)
Liver only Transplant [Number; unit: participants]
  Liver Only | 71 | 68 | 139
  Liver Plus Kidney | 11 | 14 | 25
Hepatitis C positive [Number; unit: participants]
  Hepatitis C Positive | 36 | 32 | 68
  Hepatitis C Negative | 46 | 50 | 96

OUTCOME MEASURES:

1. Primary Outcome: Rejection of Liver Transplant
Description: Liver transplant rejection determined by either biopsy or clinical criteria (>2x transaminases, clinical decision, treatment with high dose steroids and other anti-rejection medications
Time Frame: within 1 year of transplantation
Population: Patients undergoing liver transplant
Measure: Number; unit: participants
Arm/Group | 140 Group | 180 Group
Number analyzed (Participants) | 82 | 82
participants | 17 | 20
Statistical Analysis 1: Comparison: 140 Group vs 180 Group; Test type: Superiority or Other; p = 0.709, Chi-squared, Corrected

2. Secondary Outcome: Hypoglycemia
Description: Participants experiencing hypoglycemia (glucose < 70 mg/dL) within the first 3- days following transplantation
Time Frame: Within first 3 days following transplantation
Population: Patients having liver transplant
Measure: Number; unit: participants
Arm/Group | 140 Group | 180 Group
Number analyzed (Participants) | 82 | 82
participants | 27 | 10
Statistical Analysis 1: Comparison: 140 Group vs 180 Group; Test type: Superiority or Other; p = 0.003, Chi-squared, Corrected

3. Secondary Outcome: Infection Rates
Time Frame: Within 1 year following transplantation
Population: patients having had liver transplants
Measure: Number; unit: participants
Arm/Group | 140 Group | 180 Group
Number analyzed (Participants) | 82 | 82
participants | 35 | 54
Statistical Analysis 1: Comparison: 140 Group vs 180 Group; Test type: Superiority or Other; p = 0.0046, Chi-squared, Corrected

4. Secondary Outcome: Rehospitalization Rates
Time Frame: Within 1 year following transplantation
Population: patients undergoing liver transplant
Measure: Number; unit: participants
Arm/Group | 140 Group | 180 Group
Number analyzed (Participants) | 82 | 82
participants | 48 | 51
Statistical Analysis 1: Comparison: 140 Group vs 180 Group; Test type: Superiority or Other; p = 0.75, Chi-squared, Corrected

5. Secondary Outcome: Overall Graft Survival at 1 Year
Time Frame: 1 year following transplantation
Measure: Number; unit: participants
Arm/Group | 140 Group | 180 Group
Number analyzed (Participants) | 82 | 82
participants | 77 | 74
Statistical Analysis 1: Comparison: 140 Group vs 180 Group; Test type: Superiority or Other; p = 0.56, Chi-squared, Corrected

6. Secondary Outcome: Death Within 1 Year
Description: Death following liver transplant between 1 day and 1 year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | 140 Group | 180 Group
Number analyzed (Participants) | 82 | 82
participants | 5 | 7
Statistical Analysis 1: Comparison: 140 Group vs 180 Group; Test type: Superiority or Other; p = 0.77, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 1st 30 days following transplant. This is the time of the insulin/glucose intervention
Description: the major adverse event of the intervention was hypoglycemia, which is described in outcomes. There were no adverse sequelae of any of the hypoglycemic events
Arm/Group | 140 Group | 180 Group
Serious Adverse Events (participants affected / at risk) | 53/82 | 56/82
Other Adverse Events (participants affected / at risk) | 40/82 | 62/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 140 Group (N=82) | 180 Group (N=82)
death within 1 year of transplant (Hepatobiliary disorders) | 5 (5) | 5 (5) — Deaths occurring within one year of transplant
Readmission within one year (Hepatobiliary disorders) | 48 (48) | 51 (51) — Hospital readmission within one year
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 140 Group (N=82) | 180 Group (N=82)
Infections within one year of transplant (Infections and infestations) | 35 (35) | 54 (54) — Infection in any organ within one year of transplant
Liver Graft Failure within 1 year of transplant (Hepatobiliary disorders) | 5 (5) | 8 (8) — Failure of the Liver graft within 1 year of transplant

LIMITATIONS AND CAVEATS:
Single-center study with experienced nurses, glucose management service and endocrinologists. May not be applicable to other care settings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No